CLINICAL TRIAL: NCT04935879
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Safety and Efficacy of Inclacumab in Participants With Sickle Cell Disease Experiencing Vaso-occlusive Crises
Brief Title: A Study to Assess the Safety and Efficacy of Inclacumab in Participants With Sickle Cell Disease Experiencing Vaso-occlusive Crises
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT2104-131; 2020-005286-13 (EudraCT Number); C5361001 (Other: Alias Study Number)
Record Dates: First submitted 2021-05-26; First posted 2021-06-23 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Pain Episode in Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: blood disorders; hemoglobin; red blood cells; sickle-like shape; mutation in hemoglobin gene; sickle-cell trait; sickle-cell crisis; Sickle Cell Disease; SCD; Vaso-occlusive Crises; VOC; SCA; RBCs
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hematologic Diseases; Sickle Cell Trait | interventions — inclacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- inclacumab, 30 mg/kg (Experimental): Participants will receive inclacumab 30 mg/kg administered IV every 12 weeks
  Interventions: Drug: Inclacumab
- placebo (Placebo Comparator): Participants will receive placebo administered IV every 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclacumab — Inclacumab will be supplied in single use 10 mL vials at a concentration of 50 mg/mL. One vial contains 500 mg of inclacumab. This is a liquid concentrate for IV infusion.
  Arms: inclacumab, 30 mg/kg
Drug: Placebo — Placebo will be supplied in single use 10 mL vials containing the same ingredients without the active drug. Placebo will be prepared as a liquid concentrate for IV infusion and administered in the same manner as active study drug
  Arms: placebo

SUMMARY:
This Phase 3 study will assess the safety and efficacy of inclacumab, a P-selectin inhibitor, in reducing the frequency of vaso-occlusive crises (VOCs) in approximately 240 adult and adolescent participants (≥ 12 years of age) with sickle cell disease (SCD). Participants will be randomized to receive inclacumab or placebo.

DETAILED DESCRIPTION:
Eligible participants will be administered inclacumab or placebo intravenous (IV) every 12 weeks.

The total duration of treatment for each participant will be 48 weeks.

Participants that complete the study through Week 48 will be provided the opportunity to enroll in an open-label extension (OLE) study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a confirmed diagnosis of SCD (HbSS, HbSC, HbSB0 thalassemia, or HbSB+ thalassemia genotype).

   Documentation of SCD genotype is required and may be based on documented history of laboratory testing or confirmed by laboratory testing during Screening.
2. Participant is male or female, ≥ 12 years of age at the time of informed consent.
3. Participant has experienced between 2 and 10 VOCs within the 12 months prior to the Screening Visit as determined by documented medical history. A prior VOC is defined as an acute episode of pain which:

   * Has no medically determined cause other than a vaso-occlusive event, and
   * Results in a visit to a medical facility (hospital, emergency department, urgent care center, outpatient clinic, or infusion center) or results in a remote contact with a healthcare provider; and
   * Requires parenteral narcotic agents, parenteral nonsteroidal anti- inflammatory drugs (NSAIDs), or an increase in treatment with oral narcotics.
4. Participants receiving erythropoiesis-stimulating agents (ESA, e.g., erythropoietin [EPO]) must be on a stable dose for at least 90 days prior to the Screening Visit and expected to continue with the stabilized regimen throughout the course of the study.
5. Participants receiving hydroxyurea (HU), L-glutamine, or voxelotor (Oxbryta®) must be on a stable dose for at least 30 days prior to the Screening Visit and expected to continue with the stabilized regimen throughout the course of the study.

Exclusion Criteria:

1. Participant is receiving regularly scheduled red blood cell (RBC) transfusion therapy (also termed chronic, prophylactic, or preventative transfusion).
2. Participant is taking or has received crizanlizumab (ADAKVEO®) within 90 days prior to the Screening Visit
3. Participant weighs > 133 kg (292 lbs.).

Other protocol-defined Inclusion/Exclusion may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (58):
- United States (22):
  - University of South Alabama Children's and Women's Hospital, Mobile, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - University of South Alabama Strada Patient Care Center, Mobile, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC Irvine Health, Orange, California
  - UCI Center for clinical research, Orange, California
  - Uconn Health/Uconn John Dempsey Hospital/Neag Comprehensive Cancer Center/New England Sickle Cell, Farmington, Connecticut
  - Hospital Pharmacy Services- Investigational Drug Services, Chicago, Illinois
  - Rush University Medical Center Investigator Pharmacy, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Clinical Research Center (CRC), Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System(UI Health), Chicago, Illinois
  - Dana-Farber Cancer Institute IDS Pharmacy, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospitals - Michigan Medicine, Ann Arbor, Michigan
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - DUMC Investigational Drug Services Pharmacy, Durham, North Carolina
  - McGovern Medical School/Health Science Center Houston, Houston, Texas
  - Memorial Hermann - TMC Investigational Drugs, IDS Pharmacy, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center - Clinical Research Unit (CRU), Houston, Texas
  - UT Physicians Comprehensive Sickle Cell Clinic, Houston, Texas
- Brazil (9):
  - Instituto D'Or de Pesquisa e Ensino - Hospital São Rafael, Salvador, Estado de Bahia
  - Multihemo Serviços Médicos S/A, Recife, Pernambuco
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto Estadual de Hematologia Arthur Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Hospital Samaritano Higienópolis/Esho Empresa De Servicos Hospitalares S.A, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo
  - CEPEC-Centro de Pesquisa Clinica, São Paulo
- Colombia (2):
  - Clinica de la Costa Ltda., Barranquilla, Atlántico
  - Sociedad de Oncologia y hematologia del Cesar S.A.S., Valledupar, Cesar Department
- Egypt (2):
  - Faculty of Medicine Cairo University, Cairo
  - AinShams University Hospital, Cairo
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Institut Universitaire du Cancer de Toulouse-Oncopole, Toulouse
- Kenya (5):
  - KEMRI/CRDR, Siaya, KEMRI Clinical Research Annex, Kisumu, Siaya County
  - International Cancer Institute, Eldoret
  - Gertrude's Children Hospital, Nairobi
  - Kenya Medical Research Institute- Center for Respiratory Disease Research, Nairobi
  - Strathmore University Medical Center - Center for Research in Therapeutic Sciences(CREATES), Nairobi
- Lebanon (2):
  - American University of Beirut Medical Center, Hamra, Beyrouth
  - Nini Hospital, Tripoli, North Lebanon
- Nigeria (8):
  - University of Calabar Teaching Hospital, Calabar, Cross River State
  - National Hospital Abuja, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Gwagwalada, Federal Capital Territory
  - Ahmadu Bello University Teaching Hospital, Zaria, Kaduna State
  - University of Nigeria Teaching Hospital, Enugu
  - Barau Dikko Teaching Hospital/Kaduna State University, Kaduna
  - Aminu Kano Teaching Hospital, Kano
  - Department of Pediatrics, College of Medicine, Lagos University Teaching Hospital, Lagos
- Sultan َQaboos University Hospital, Muscat, Oman
- Prince Mohammed bin Nasser Hospital, Jizan, Southern, Saudi Arabia
- NIMR-Mbeya Medical Research Center, Mbeya, Tanzania
- Turkey (Türkiye) (3):
  - Mersin Universitesi Tip Fakultesi Saglik Arastirma ve Uygulama Merkezi Hastanesi, Yenişehir, Mersin
  - Baskent University Hospital, Adana, Yuregir
  - Acibadem Adana Hastanesi Cocuk Hematoloji Onkoloji, Adana

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT2104-131

RESULTS

PARTICIPANT FLOW:
Groups:
- Inclacumab: Participants with sickle cell disease (SCD) were randomized to receive inclacumab at a dose of 30 milligram/kilogram (mg/kg) intravenously (IV) on Day 1 and once every 12 weeks (Q12W) on Weeks 12, 24 and 36. Participants were followed up till Week 48 and was part of "48-Week Treatment Period". Participants at Week 48 had a choice to either enter an open-label extension (OLE) study (under a separate protocol) to receive inclacumab or were followed up for another 12 weeks i.e. Week 60.
- Placebo: Participants with SCD were randomized to receive placebo matched to inclacumab IV on Day 1 and Q12W on Weeks 12, 24 and 36. Participants were followed up till Week 48 and was part of "48-Week Treatment Period". Participants at Week 48 had a choice to either enter an OLE study (under a separate protocol) to receive inclacumab or were followed up for another 12 weeks i.e. Week 60.
Period: Overall Study
Arm/Group | Inclacumab | Placebo
Started | 119 | 122
Treated | 118 | 121
Completed | 103 | 108
Not Completed | 16 | 14
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 2 | 3
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- Inclacumab: Participants with SCD were randomized to receive inclacumab at a dose of 30 mg/kg IV on Day 1 and Q12W on Weeks 12, 24 and 36. Participants were followed up till Week 48 and was part of "48-Week Treatment Period". Participants at Week 48 had a choice to either enter an OLE study (under a separate protocol) to receive inclacumab or were followed up for another 12 weeks i.e. Week 60.
- Total: Total of all reporting groups
Arm/Group | Inclacumab | Placebo | Total
Number analyzed (Participants) | 119 | 122 | 241
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.0 (7.14) | 24.6 (8.34) | 24.8 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 63 | 127
  Male | 55 | 59 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 19 | 37
  Not Hispanic or Latino | 92 | 102 | 194
  Unknown or Not Reported | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African | 63 | 58 | 121
  Race: American Indian or Alaska Native | 3 | 2 | 5
  Race: Arab | 1 | 2 | 3
  Race: Black or African American | 16 | 24 | 40
  Race: Middle Eastern | 1 | 0 | 1
  Race: Other | 2 | 1 | 3
  Race: Multiracial | 22 | 25 | 47
  Race: Not Reported | 4 | 0 | 4
  Race: White | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Rate of Vaso-occlusive Crises (VOCs) [Adjudicated] Through Week 48
Description: A VOC was defined as an acute episode of pain that: had no medically determined cause other than a vaso-occlusive event; resulted in a visit to a medical facility (hospitalization, emergency department, urgent care center, outpatient clinic, or infusion center), or resulted in a remote contact with a healthcare provider and required parenteral narcotic agents, parenteral nonsteroidal anti-inflammatory drugs (NSAIDs), or an increase in treatment with oral narcotics. The rate of VOC was defined as number of VOC events per 48 weeks and presented in this outcome measure.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Events per 48 weeks
Groups:
- Inclacumab: Participants with SCD were randomized to receive inclacumab at a dose of 30 mg/kg IV on Day 1 and Q12W on Weeks 12, 24 and 36.Participants were followed up till Week 48 and was part of "48-Week Treatment Period". Participants at Week 48 had a choice to either enter an OLE study (under a separate protocol) to receive inclacumab or were followed up for another 12 weeks i.e. Week 60.
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Events per 48 weeks | 1.49 [1.22 to 1.83] | 1.58 [1.30 to 1.93]
Statistical Analysis 1: Comparison: Inclacumab vs Placebo; Adjusted rates are based on estimate from a negative binomial model with the independent variable of treatment group (inclacumab, placebo) and adjusted for baseline hydroxyurea (HU) use (yes, no), number of VOCs in 12 months prior to screening visit (2-4, 5-10), and geographic region (North America, sub-Saharan Africa, Europe/rest of world); Test type: Superiority; p = 0.6967, Negative binomial regression model; Rate ratio = 0.95, 95% CI 2-sided [0.71 to 1.25] — Rate ratio = Ratio of rate of VOC for inclacumab group to placebo group

2. Secondary Outcome: Time to First VOC Through Week 48
Description: A VOC was defined as an acute episode of pain that: had no medically determined cause other than a vaso-occlusive event; resulted in a visit to a medical facility (hospitalization, emergency department, urgent care center, outpatient clinic, or infusion center), or resulted in a remote contact with a healthcare provider and required parenteral narcotic agents, parenteral NSAIDs, or an increase in treatment with oral narcotics. Time to first VOC was the time between randomization date and onset date of first VOC event during 48 weeks. Kaplan-Meier method was used for estimation.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Weeks | 28.7 [15.7 to 43.1] | 21.6 [17.3 to 28.7]
Statistical Analysis 1: Comparison: Inclacumab vs Placebo; Analysis was stratified by baseline HU use (yes, no), number of VOCs in 12 months prior to screening visit (2-4, 5-10), and geographic region (North America, sub-Saharan Africa, Europe/rest of world); Test type: Superiority; p = 0.4298, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.63 to 1.22]

3. Secondary Outcome: Time to Second VOC Through Week 48
Description: A VOC was defined as an acute episode of pain that: had no medically determined cause other than a vaso-occlusive event; resulted in a visit to a medical facility (hospitalization, emergency department, urgent care center, outpatient clinic, or infusion center), or resulted in a remote contact with a healthcare provider and required parenteral narcotic agents, parenteral NSAIDs, or an increase in treatment with oral narcotics. Time to second VOC was the time between randomization date and onset date of second VOC event during 48 weeks. Kaplan-Meier method was used for estimation.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Weeks | NA [NA to NA] — Median, upper and lower limit of 95% confidence interval (CI) was not estimated due to insufficient number of participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI was not estimated due to insufficient number of participants with events.

4. Secondary Outcome: Percentage of Participants With no VOCs Through Week 48
Description: A VOC was defined as an acute episode of pain that: had no medically determined cause other than a vaso-occlusive event; resulted in a visit to a medical facility (hospitalization, emergency department, urgent care center, outpatient clinic, or infusion center), or resulted in a remote contact with a healthcare provider and required parenteral narcotic agents, parenteral NSAIDs, or an increase in treatment with oral narcotics. Participants without an observed VOC who discontinued the study prior to the end of the 48-week treatment period were assumed to had experienced at least one VOC.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Percentage of participants | 36.0 [27.1 to 45.0] | 25.7 [17.7 to 33.7]
Statistical Analysis 1: Comparison: Inclacumab vs Placebo; Cochran-Mantel-Haenszel (CMH) test stratified by baseline HU use (yes, no), number of VOCs in the 12 months prior to study entry (2-4, 5-10), and geographic region (North America, sub-Saharan Africa, Europe/rest of world); Test type: Superiority; p = 0.0912, Cochran-Mantel-Haenszel; Difference in Percentage = 10.3, 95% CI 2-sided [-1.6 to 22.2]

5. Secondary Outcome: Rate of VOCs Required Admission to a Healthcare Facility and Treatment With Parenteral Pain Medication [Adjudicated] Through Week 48
Description: A VOC that required admission to a healthcare facility and treatment with parenteral pain medication where admission included: a hospital admission or an admission to an emergency room, observation unit, or infusion center for >= 12 hours, or 2 visits to an emergency room, observation unit, or infusion center over a 72-hour period. The rate of VOC was defined as number of VOC events per 48 weeks; rate of VOCs which required admission to a healthcare facility and treatment with parenteral pain medication is presented in this outcome measure.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Events per 48 weeks
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Events per 48 weeks | 0.85 [0.65 to 1.10] | 0.83 [0.64 to 1.08]
Statistical Analysis 1: Comparison: Inclacumab vs Placebo; Adjusted rates are based on estimate from a negative binomial model with the independent variable of treatment group (inclacumab, placebo) and adjusted for baseline HU use (yes, no), number of VOCs in the 12 months prior to screening visit (2-4, 5-10), and geographic region (North America, sub-Saharan Africa, Europe/rest of the world); Test type: Superiority; p = 0.9246, Negative binomial regression model; Rate Ratio = 1.02, 95% CI 2-sided [0.71 to 1.47] — Rate ratio = Ratio of rate of VOC for inclacumab group to placebo group

6. Secondary Outcome: Rate of Inpatient Hospitalization Days for a VOC Through Week 48
Description: A VOC was defined as an acute episode of pain that: had no medically determined cause other than a vaso-occlusive event; resulted in a visit to a medical facility hospitalization. For each VOC event requiring inpatient hospitalization (regardless of treatment received) during the 48-week, the number of days hospitalized were determined based on the hospital admission and discharge dates. The rate of inpatient hospitalization days was defined as number of inpatient hospitalization days for a VOC per 48 weeks and presented in this outcome measure.
Time Frame: Randomization (Day 1) up to Week 48
Population: The ITT population included all randomized participants.
Measure: Number (95% Confidence Interval); unit: Hospitalization days per 48 weeks
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 119 | 122
Hospitalization days per 48 weeks | 4.96 [3.05 to 8.07] | 5.37 [3.34 to 8.62]
Statistical Analysis 1: Comparison: Inclacumab vs Placebo; Adjusted rates are based on estimate from a negative binomial model with the independent variable of treatment group (inclacumab, placebo) and adjusted for baseline HU use (yes, no), number of VOCs in 12 months prior to screening visit (2-4, 5-10), and geographic region (North America, sub-Saharan Africa, Europe/rest of world); Test type: Superiority; p = 0.8263, Negative binomial regression model; Rate ratio = 0.92, 95% CI 2-sided [0.46 to 1.87] — Rate ratio = Ratio of rate of VOC for inclacumab group to placebo group

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product during the course of a clinical investigation. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of an investigational product, whether or not thought to be related to the investigational product. A TEAE was defined as an AE with an onset after the initiation of dosing for the first dose of study drug. A serious adverse events (SAE) or serious suspected adverse reaction is an AE or suspected adverse reaction that, at any dose, in the view of the either the investigator or sponsor, results in any of the following outcomes: death, life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization and congenital anomaly/birth defect. AEs included both serious and all non-SAEs.
Time Frame: Day 1 up to Week 60 (12 week of follow-up post Week 48)
Population: Safety population included randomized participants who received treatment with study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Inclacumab | Placebo
Number analyzed (Participants) | 118 | 121
Participants | 87 [3.05 to 8.07] | 97 [3.34 to 8.62]

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 60 (12 week of follow-up post Week 48)
Description: Same event may appear as both non-SAE and SAE, but what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. The safety population included randomized participants who received treatment with study drug.
Arm/Group | Inclacumab | Placebo
All-Cause Mortality (participants affected / at risk) | 3/118 | 2/121
Serious Adverse Events (participants affected / at risk) | 23/118 | 27/121
Other Adverse Events (participants affected / at risk) | 83/118 | 90/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclacumab (N=118) | Placebo (N=121)
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Haemolysis (Blood and lymphatic system disorders) | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Malaria (Infections and infestations) | 5 | 7
Pneumonia (Infections and infestations) | 5 | 5
Bacterial infection (Infections and infestations) | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclacumab (N=118) | Placebo (N=121)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 21 | 21
Anaemia (Blood and lymphatic system disorders) | 5 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Cor pulmonale acute (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 0
Pterygium (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 0 | 1
Retinopathy sickle cell (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Toothache (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 7 | 4
Pain (General disorders) | 6 | 5
Non-cardiac chest pain (General disorders) | 4 | 1
Fatigue (General disorders) | 3 | 2
Asthenia (General disorders) | 2 | 1
Chest pain (General disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Injury associated with device (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 1
Sluggishness (General disorders) | 0 | 1
Swelling (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Ocular icterus (Hepatobiliary disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Malaria (Infections and infestations) | 18 | 24
Nasopharyngitis (Infections and infestations) | 9 | 2
Upper respiratory tract infection (Infections and infestations) | 9 | 12
COVID-19 (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 2 | 3
Influenza (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 2 | 3
Respiratory tract infection (Infections and infestations) | 2 | 2
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 3
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 7
Vulvovaginitis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 8
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Wound sepsis (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1
Vascular access site pruritus (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Fibrin D dimer increased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
C-reactive protein (Investigations) | 1 | 0
Coagulation test abnormal (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Neutrophil count abnormal (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 1 | 0
Prothrombin time shortened (Investigations) | 1 | 0
Reticulocyte count increased (Investigations) | 1 | 1
Reticulocyte percentage increased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Neutrophil count increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperferritinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 16 | 21
Migraine (Nervous system disorders) | 2 | 1
Ageusia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Amputation stump pain (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 1 | 1
Psychogenic seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 2 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0
Penile swelling (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis alba (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 1
Flushing (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hyperaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04935879/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT04935879/SAP_002.pdf